CLINICAL TRIAL: NCT07050459
Title: A Phase I First-in-Human, Open-label, Multicenter Study to Investigate the Safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of SIM0686 in Adult Participants With Locally Advanced/Metastatic Solid Tumors
Brief Title: A Phase I Study of SIM0686 in Participants With Locally Advanced/Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SIM0686-101
Record Dates: First submitted 2025-05-27; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Locally Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SIM0686 momo Dose escalation (Experimental): Sequential cohorts of increasing dose levels of SIM0686 will be evaluated as monotherapy
  Interventions: Drug: SIM0686
- SIM0686 Corhort expansion (Experimental): Recommended Dose(s) of SIM0686 as determined from Part1 will be evaluated in select indications
  Interventions: Drug: SIM0686

INTERVENTIONS:
Drug: SIM0686 — Administered intravenously
  Arms: SIM0686 Corhort expansion
Drug: SIM0686 — Administered intravenously
  Arms: SIM0686 momo Dose escalation

SUMMARY:
This is an open-label, multicenter phase 1 study to evaluate the safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of SIM0686 in Adult Participants with Locally Advanced/Metastatic Solid Tumors

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation and signature of informed consent form;
* At least 18 years old, male, or female;
* Participants with histologically and/or cytologically confirmed locally advanced/metastatic solid tumors;
* Participants should have at least one evaluable or measurable tumor lesion (RECIST v1.1);
* Participants have failed the standard of therapy in the locally advanced/metastatic setting
* Eastern Cooperative Oncology Group (ECOG) performance score of 0 or 1;
* Expected survival ≥12 weeks;
* Adequate organ and bone marrow function;
* Availability of archival formalin-fixed, paraffin-embedded (FFPE) tumor tissue, or fresh biopsies within 6 months before first administration for evaluation of FGFR2b expression levels

Exclusion Criteria:

* Active second primary malignancies within the previous 2 years except for localized cancers that are considered to have been cured and in the opinion of the Investigator present a low risk for recurrence.
* Participant has symptomatic central nervous system (CNS) metastases, or CNS metastases requiring CNS-directed local therapy (such as radiotherapy or surgery) or corticosteroids therapy within 2 weeks of first dose of study treatment.
* Active or chronic corneal disorder, history of corneal transplantation, keratitis, keratoconjunctivitis, keratopathy, keratoconus, corneal abrasion, inflammation or ulceration, other active ocular conditions and any clinically significant corneal disease that prevents adequate monitoring of drug-induced keratopathy.
* Has a history of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids, current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging screening.
* Participant has not recovered (i.e., to Grade 1 or to baseline) from previous anticancer therapy-induced AEs.
* Has received prior therapies within the following time frames prior to the first dose of study treatment:

  1. Previous cytotoxic therapy, anticancer targeted small molecules (e.g., tyrosine kinase inhibitors) within 2 weeks.
  2. Anti-cancer antibody, immune checkpoint inhibitor or ADC within 5 half-lives or 4 weeks (whichever is shorter).
  3. Chinese medicines/herbal preparations with anticancer indication taken within 2 weeks.
  4. Radiation therapy within 4 weeks.
* Prior exposure to topoisomerase I inhibitor (TOP1i)-based antibody-drug conjugate (ADC) therapies or FGFR2b-targeted ADC therapies.
* Known human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS).
* Active or chronic hepatitis B or hepatitis C infection;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Dose escalation: Dose limited toxicity (DLT) | At the end of Cycle 1(each cycle is 21 days)
  DLTs are assessed during the DLT observation period to determine maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D).
Dose escalation phase: Adverse Events (AEs) and Serious Adverse Events (SAEs) | The whole dose escalation phase，an average of 2 years
  Adverse events will be assessed by investigator(s) according to NCI-CTCAE v5.0.
Cohort expansion phase：Overall Response Rate (ORR) | The whole Cohort expansion phase，an average of 2 years
  ORR is defined as the percentage of participants with confirmed complete response (CR) or partial response (PR) by Response Evaluations Criteria in Solid Tumors Version 1.1 (RECIST v1.1)

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Harbin Medical University Cancer Hospital, Haerbin, Heilongjiang
  - The Affiliated Cancer Hospital of Zhengzhou University & Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Tianyinshan Hospital, Nanjing, Jiangsu
  - Cancer Hospital of Shandong First Medical University（Shandong Cancer Hospital&Institute）, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai Gobroad Cancer Hospital, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality